CLINICAL TRIAL: NCT01934387
Title: Increasing Osteoporosis Awareness With Fracture Risk Assessments and Management Among Geriatric Health Examination Recipients at National Taiwan University Hospital
Brief Title: Geriatric Health Exam Osteoporosis Screening
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201205110RIC
Record Dates: First submitted 2013-07-03; First posted 2013-09-04 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Osteoporosis; Accidental Falls; Fracture
Keywords: World Health Organization Fracture Risk Assessment Tool; Osteoporosis; Aged; Prevention; Fracture; FRAX
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
BACKGROUND: The World Health Organization Fracture Risk Assessment Tool (WHO FRAX®) Taiwanese calculator is freely available on line to help osteoporosis management. However, its clinical utility for improving osteoporosis awareness and patient acceptance has not been validated in Taiwanese population.

OBJECTIVES: This 11-month FRAX® based screening and referral program enrolling older adults participating in the geriatric health examinations (GHEs) at the National Taiwan University Hospital (NTUH) aiming at determine the patient acceptance of the tool and the program and to improve patient awareness in osteoporosis. The second aim is to look for the recommendations from the participating physicians to improve the FRAX® -based osteoporosis management model.

METHODS: The NTUH GHE program is a two stage process to serve 3,000 older adults collecting annually from Mar. to Dec. Subjects will be enrolled to the current study at the stage 1 GHE visits after informed consent. Baseline questionnaires including the FRAX® tools will be distributed and expected to be returned at the stage 2 visits. Research assistants will calculate the 10-year predicted fracture risks for the participants during the waiting periods and present the numbers to the GHE physicians. High risks individuals will be referred to general geriatric clinic for further managements. All participants will be provided with osteoporosis and fracture educational material. Patient acceptance and awareness will be assessed. The study is to be started from Feb., to Oct., 2013 to enroll roughly 1,800 older adults assuming refusal rate about 40%.

Qualitative interviews will be used to obtain recommendations from study geriatricians in Jul., 2013 to optimize the FRAX® based screening and management model.

DETAILED DESCRIPTION:
ANTICIPATED RESULTS:

To estimate the 10 year fracture risks for GHE participants. To understand the acceptance of this FRAX® based model from GHE participants and the impacts on patient osteoporosis awareness.

To calculate the economic benefits of this model on geriatric outpatient service.

To obtain recommendations from study geriatricians to optimize the FRAX® based model for further disseminations.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the NTUH GHE program
* Can complete the study questionnaire
* Willingness to join in the researchers

Exclusion Criteria:

* NA

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Adults visitng geraitric health exam clinics.
Sampling Method: Non-Probability Sample
Enrollment: 1319 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Percentages of elderly transfer to geriatric department | 11-month
  The study expected to collect 1,800 cases that using the assessment tool (FRAX) for osteoporosis screening. The primary outcomes were 10-year probability of major osteoporotic fracture and 10-year probability of hip fracture.Investigators want to know what the percentages of elderly in high risk need to be transfer to geriatric department for further treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan